CLINICAL TRIAL: NCT02280967
Title: Prevention of Human Papillomavirus (HPV) Associated Cancer by Intervention Studies in Teenagers Attending School Health
Brief Title: Prevention of HPV in the School Health Service
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Swedish Cancer Society (Other); Uppsala-Örebro Regional Research Council (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RFR-387561
Record Dates: First submitted 2014-10-21; First posted 2014-11-03 (Estimated); Last update posted 2017-09-05 (Actual); Status verified 2017-09

CONDITIONS: Human Papillomavirus; Cervix Cancer
Keywords: Adolescent; Attitude; Condom; Human Papillomavirus Vaccines; Primary prevention; School Health
MeSH Terms: conditions — Uterine Cervical Neoplasms; Behavior

STUDY DESIGN:
Masking Description: Open label
Oversight: Data Monitoring Committee: No

ARMS (2):
- Education about HPV by school nurse (Experimental): The educational intervention consists of education about HPV and a special designed leaflet and self-reported questionnaires. The educational intervention is included in the regular health interview with the school nurse (scheduled for about one hour) and includes information about HPV; facts about the virus, transmission, what it can cause and prevention (i.e. safe sex with condom use and HPV vaccination), facts about HPV vaccine and the importance of attending future cervical cancer screening controls. Students complete questionnaires before the health interview at baseline and after three months. A follow-up with parts of the boys will be performed with qualitative interviews. Participants (n=40)
  Interventions: Behavioral: Education about HPV by school nurse
- Control group 1 (No Intervention): Students allocated to control group 1 receives standard treatment, the regular health interview with the school nurse. Students complete questionnaires before the health interview at baseline and after three months (n=400).

INTERVENTIONS:
Behavioral: Education about HPV by school nurse — Information about prevention of HPV among adolescents aged 16 at time for the regular health interview with the school nurse.
  Arms: Education about HPV by school nurse

SUMMARY:
The last ten years sexually transmitted infections (STI) have substantially increased among adolescents. STI can lead to individual suffering and have a negative effect on the future reproductive health and also increase the need for health care, thus it is important to reduce the number of STIs. HPV vaccination is included in the school-based vaccination program since 2012, a catch-up vaccination is offered to older girls and young women aged 13-25. School nurses have a key role regarding information about HPV and HPV vaccine, and the school-based vaccination program has a substantial higher coverage rate. Knowledge is an important factor associated with attitude to preventive methods against HPV. In previous studies the results indicate that young people have low awareness of HPV and the HPV vaccine. Interventions can decrease sexual risk taking and influence the intention to receive HPV vaccination and increase the use of condom.

The aim of this study is to increase primary prevention of human papillomavirus (HPV) by promoting HPV vaccination and increase condom use among upper secondary students. The aim is also to increase the knowledge about HPV, risk and prevention.

ELIGIBILITY:
Inclusion Criteria:

* First year students in upper secondary school who visit the school nurse for the regular health interview.
* Master Swedish in speech and writing.

Exclusion Criteria:

* Students with cognitive disabilities.

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 832 (Actual)
Dates: Start 2014-01; Primary Completion 2017-08 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Intention to use condom if new partner | Change from Baseline Intention at 3 months
  Intention to use condom if new partner measured by questionnaire, five-point Likert scale ranging from "totally agree" to "totally disagree".
Intention to use condom if new partner | Change from Baseline Intention at 12 months
  Intention to use condom if new partner measured by questionnaire, five-point Likert scale ranging from "totally agree" to "totally disagree".
Intention to use condom if new partner | Change from Baseline Intention at 24 months
  Intention to use condom if new partner measured by questionnaire, five-point Likert scale ranging from "totally agree" to "totally disagree".
Attitude to prevention about HPV | Change from Baseline Attitude at 3 months
  Attitude to HPV vaccine. Intention to be vaccinated against HPV. Condom use and intention to attend future cervical cancer screening programmes. Measured by questionnaire, five-point Likert scale ranging from "totally agree" to "totally disagree".
Attitude to prevention about HPV | Change from Baseline Attitude at 12 months
  Attitude to HPV vaccine. Intention to be vaccinated against HPV. Condom use and intention to attend future cervical cancer screening programmes. Measured by questionnaire, five-point Likert scale ranging from "totally agree" to "totally disagree".
Attitude to prevention about HPV | Change from Baseline Attitude at 24 months
  Attitude to HPV vaccine. Intention to be vaccinated against HPV. Condom use and intention to attend future cervical cancer screening programmes. Measured by questionnaire, five-point Likert scale ranging from "totally agree" to "totally disagree".

SECONDARY OUTCOMES:
Behavioural outcomes: Increased HPV vaccination and increased condom use. | Change from Baseline Behaviour at 3 months.
  Measured by questionnaire. Vaccinated against HPV? Condom use at last sexual intercourse?
Behavioural outcomes: Increased HPV vaccination and increased condom use. | Change from Baseline Behaviour at 12 months.
  Measured by questionnaire. Vaccinated against HPV? Condom use at last sexual intercourse?
Behavioural outcomes: Increased HPV vaccination and increased condom use. | Change from Baseline Behaviour at 24 months.
  Measured by questionnaire. Vaccinated against HPV? Condom use at last sexual intercourse?

OTHER OUTCOMES:
Knowledge about HPV | Change from Baseline Knowledge at 3 months
  Knowledge about HPV measured by questionnaire. (Facts about the virus, transmission, what HPV can cause. Heard of HPV vaccine?)
Knowledge about HPV | Change from Baseline Knowledge at 12 months
  Knowledge about HPV measured by questionnaire. (Facts about the virus, transmission, what HPV can cause. Heard of HPV vaccine?)
Knowledge about HPV | Change from Baseline Knowledge at 24 months
  Knowledge about HPV measured by questionnaire. (Facts about the virus, transmission, what HPV can cause. Heard of HPV vaccine?)

CONTACTS AND LOCATIONS:
Overall Officials: Tanja Tydén, Professor, Study Director — Uppsala University
Locations (1):
- Uppsala University, Public Health and Caring Sciences, Uppsala, Sweden

REFERENCES:
- [Background] Shepherd J, Kavanagh J, Picot J, Cooper K, Harden A, Barnett-Page E, Jones J, Clegg A, Hartwell D, Frampton GK, Price A. The effectiveness and cost-effectiveness of behavioural interventions for the prevention of sexually transmitted infections in young people aged 13-19: a systematic review and economic evaluation. Health Technol Assess. 2010 Feb;14(7):1-206, iii-iv. doi: 10.3310/hta14070. PMID 20178696
- [Background] Fu LY, Bonhomme LA, Cooper SC, Joseph JG, Zimet GD. Educational interventions to increase HPV vaccination acceptance: a systematic review. Vaccine. 2014 Apr 7;32(17):1901-20. doi: 10.1016/j.vaccine.2014.01.091. Epub 2014 Feb 14. PMID 24530401
- [Result] Danielsson M, Berglund T, Forsberg M, Larsson M, Rogala C, Tyden T. Sexual and reproductive health: Health in Sweden: The National Public Health Report 2012. Chapter 9. Scand J Public Health. 2012 Dec;40(9 Suppl):176-96. doi: 10.1177/1403494812459600. No abstract available. PMID 23238407
- [Result] Gottvall M, Grandahl M, Hoglund AT, Larsson M, Stenhammar C, Andrae B, Tyden T. Trust versus concerns-how parents reason when they accept HPV vaccination for their young daughter. Ups J Med Sci. 2013 Nov;118(4):263-70. doi: 10.3109/03009734.2013.809039. Epub 2013 Jun 19. PMID 23777602
- [Result] Grandahl M, Oscarsson M, Stenhammar C, Neveus T, Westerling R, Tyden T. Not the right time: why parents refuse to let their daughters have the human papillomavirus vaccination. Acta Paediatr. 2014 Apr;103(4):436-41. doi: 10.1111/apa.12545. Epub 2014 Jan 8. PMID 24460679
- [Result] Grandahl M, Tyden T, Rosenblad A, Oscarsson M, Neveus T, Stenhammar C. School nurses' attitudes and experiences regarding the human papillomavirus vaccination programme in Sweden: a population-based survey. BMC Public Health. 2014 May 31;14:540. doi: 10.1186/1471-2458-14-540. PMID 24886332
- [Result] Shepherd JP, Frampton GK, Harris P. Interventions for encouraging sexual behaviours intended to prevent cervical cancer. Cochrane Database Syst Rev. 2011 Apr 13;2011(4):CD001035. doi: 10.1002/14651858.CD001035.pub2. PMID 21491379
- [Derived] Grandahl M, Rosenblad A, Stenhammar C, Tyden T, Westerling R, Larsson M, Oscarsson M, Andrae B, Dalianis T, Neveus T. School-based intervention for the prevention of HPV among adolescents: a cluster randomised controlled study. BMJ Open. 2016 Jan 27;6(1):e009875. doi: 10.1136/bmjopen-2015-009875. PMID 26817639